CLINICAL TRIAL: NCT06182319
Title: The Use of Nasogastric Tubes And Water-Soluble Contrast In The Management Of Small Bowel Obstruction: A Feasibility Study
Brief Title: Optimizing Treatment of Adhesive Small Bowel Obstruction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edward Harry Livingston, Professor of Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-001055
Record Dates: First submitted 2023-11-30; First posted 2023-12-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: nasogastric tube (NGT); water-soluble contrast (WSC); Adhesion-related SBO (aSBO); Small bowel obstruction (SBO)
MeSH Terms: interventions — Diatrizoate Meglumine; Sodium Chloride; Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: Patients will be allocated into 3 groups: One treated without NG tubes. The other 2 groups will have an NG tube and be randomized into treatment with water-soluble contrast or saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SBO treated without NG tube (Experimental): Patients who decline NG intubation will be enrolled in the trial, followed prospectively and have the same outcome measures as are acquired in the other study arms.
  Interventions: Procedure: SBO Treatment Without NG Tubes
- SBO treated with NG tube and Water-Soluble Contrast (WSC) (Experimental): Patients who select NG tube treatment will be randomized into experimental and control groups. The experimental groups will have 100 cc of WSC administered in the NG tube within 2 hours of NG tube placement.
  Interventions: Drug: Gastrografin
- SBO Treated with NG tube and Placebo (Placebo Comparator): The control group will have 100cc of saline administered via the NG tube within 2 hours of NG tube placement.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Gastrografin — Administration of WSC (Gastrografin) 2 hours after placement of NGT.
  Arms: SBO treated with NG tube and Water-Soluble Contrast (WSC)
Drug: Saline — Administration of Saline 2 hours after placement of NGT.
  Arms: SBO Treated with NG tube and Placebo
Procedure: SBO Treatment Without NG Tubes — Patients who decline to have NG tubes placed will be enrolled and followed with the same outcomes protocol as the other patients in the trial
  Arms: SBO treated without NG tube

SUMMARY:
Small bowel obstruction (SBO) is one of the most common causes of serious gastrointestinal disease in the US. Adhesion-related SBO (aSBO) is usually treated by the placement of a nasogastric tube (NGT) to decompress the stomach, administration of intravenous (IV) fluids and observation by a surgical team.

The purpose of this feasibility study is to determine the potential for implementation of treatment protocols for aSBO and determine the feasibility of randomizing patients with aSBO to receive or not receive NGTs or water-soluble contrast (WSC). The investigators will also determine the ability to measure HRQOL as a main outcome for the treatment of aSBO. The studies outlined in this research program intend to address gaps in knowledge about how to determine who benefits from NGT placement, who can be managed without them, how to objectively determine when a bowel obstruction has resolved, how to reintroduce feeding to patients with aSBO, what criteria should be used for hospital discharge and what role cathartics such as WSC contrast have in the management of aSBO.

This feasibility study will enroll a limited number of patients (n=40) who will be followed for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Documentation of aSBO as evidenced by one or more clinical features meeting the following criteria: Nausea, emesis, abdominal pain, distended abdomen CT evidence of aSBO

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
3. Unstable angina or recent myocardial infarction (MI)/stroke within 6 months
4. Nonadhesive SBO

   1. Paralytic Ileus
   2. Incarcerated hernia
   3. Fecal impaction
   4. Intra-abdominal malignancy Early aSBO within 4 weeks of a prior abdominal operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS®)-29 | The measure will be obtained at baseline when a diagnosis of aSBO is made, at hospital day 1, the day after an NGT is removed, the day a patient is discharged from the hospital and at 30 days after discharge.
  Quality of life will be assessed using the PROMIS-29 HRQOL instrument. The survey uses multiple response formats. A total score provides an index of HRQOL, with higher scores on a scale of 0-100 reflecting better HRQOL.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, David Geffen School of Medicine, Los Angeles, California, United States

REFERENCES:
- See also: The Effect of Hyperosmolar Water-Soluble Contrast for the Management of Adhesive Small Bowel Obstruction: A Systematic Review and Meta-Analysis — http://pubmed.ncbi.nlm.nih.gov/35837888/
- See also: Management of small bowel obstruction and systematic review of treatment without nasogastric tube decompression — http://pubmed.ncbi.nlm.nih.gov/36992798/